CLINICAL TRIAL: NCT04578808
Title: Unruptured Cerebral Aneurysm: Prediction of Evolution
Acronym: U-CAN
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0012
Record Dates: First submitted 2020-09-09; First posted 2020-10-08 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Unruptured Intracranial Aneurysm
Keywords: Unruptured Cerebral Aneurysm; Aneurysm Prediction Growth; Unruptured Intracranial aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Unruptured intracranial aneurysms — UIA of bifurcation between 3 and 7 mm for whom a clinical and imaging follow-up without occlusion treatment was scheduled by local multidisciplinary staff will be included. Extensive clinical, biological and imaging data will be recorded during a 3 years follow-up (visits at 1 and 3 years after inclusion).

SUMMARY:
The protocol has many assets. A prospective nationwide recruitment allows for the inclusion of a large cohort of patients with UIA. It will combine accurate clinical phenotyping and comprehensive imaging with CAWE screening. Besides, it will enable to exploit metadata and to explore new pathophysiological pathways of interest by crossing clinical, genetic, biological, and imaging information.

DETAILED DESCRIPTION:
Management of small (<7mm) unruptured intracranial aneurysms (UIA) remains controversial. Previous retrospective studies have suggested that post gadolinium arterial wall enhancement (AWE) of unruptured intracranial aneurysms on MR imaging may reflect aneurysm wall instability, and hence may highlight a higher risk of UIA growth over time. This multicentric prospective cohort aims at exploring vessel wall imaging findings of UIAs with consecutive follow-up to substantiate these assumptions.The objective is to develop diagnostic and predictive tools for the risk of IA evolution. The aim is to demonstrate in clinical practice the predictive value of (AWE) for UIA growth. The growth will be determined by any modification of the UIA measurement. Both UIA growth and the UIA wall enhancement will be assessed in consensus by two expert neuroradiologists.The French prospective UCAN project is a non-interventional international wide and multicentric prospective cohort. UIA of bifurcation between 3 and 7 mm for whom a clinical and imaging follow-up without occlusion treatment was scheduled by local multidisciplinary staff will be included. Extensive clinical, biological and imaging data will be recorded during a 3 years follow-up (visits at 1 and 3 years after inclusion).

ELIGIBILITY:
Inclusion Criteria :

* Subject carrying unruptured, asymptomatic and untreated typical IA of bifurcation, measured on conventional imaging (MRI, CTA or DSA) between 3 and 7 mm of larger diameter.
* Ability to be followed-up during 3 years decided in consensus multidisciplinary gathering.
* Age > 18 years old.

Exclusion Criteria :

* A failure to obtain informed consent
* Contraindications for undergoing an MRI scan include : (heart pacemaker, a metallic foreign body (metal sliver) in their eye, or aneurysm clip in their brain, severe claustrophobia)
* Contraindications for a gadolinium contrast medium injection (:eGFR below 30 mL/min/1.73 m2, Previous or pre-existing nephrogenic systemic fibrosis, Previous anaphylactic/anaphylactoid reaction to gadolinium containing contrast agent, Acutely deteriorating renal function, Pregnancy and breast-feeding)
* A mycotic, fusiform-shaped, or dissecting IA, an IA in relation with an arteriovenous malformation
* A family history of polycystic kidney disease, Ehlers-Danlos syndrome, Marfan's syndrom, fibromuscular dysplasia, or Moya Moya disease
* Intra-cavernous UIA because the sinus cavernous that is fulfilled with venous blood precluded a reliable assessment of aneurysmal wall enhancement (AWE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruited population is composed of subjects carrying unruptured asymptomatic typical IA of bifurcation for whom a clinical, a biological and an imaging follow-up, without occlusion treatment, was scheduled by local multidisciplinary staff.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-03-15 (Estimated)

PRIMARY OUTCOMES:
The aim is to evaluate in clinical practice the predictive value of UIA wall enhancement for UIA growth. It will allow to set up a secure, efficient and personalized follow-up. | 5 years
  In order to evaluate the informative value of AWE for UIA growth, investigators will consider as primary endpoint the growth of the UIA after the complete follow-up at 3 years.
Predictive value of UIA wall enhancement for UIA growth | at 1 year
  This event could occur at any time during the follow-up if an UIA becomes symptomatic but will be systematically assessed by MRI. UIA growth will be assessed blindly and independently by two expert neuroradiologists, routinely involved in UIA management and disagreement will be solved by consensus with involvement of a third expert. UIA wall enhancement status will be defined independently by two different expert neuroradiologists, with > 5yrs experience in intracranial vessel wall imaging. Disagreement will be solved by consensus with involvement of a third expert.
Predictive value of UIA wall enhancement for UIA growth | at 3 years
  This event could occur at any time during the follow-up if an UIA becomes symptomatic but will be systematically assessed by MRI. UIA growth will be assessed blindly and independently by two expert neuroradiologists, routinely involved in UIA management and disagreement will be solved by consensus with involvement of a third expert. UIA wall enhancement status will be defined independently by two different expert neuroradiologists, with > 5yrs experience in intracranial vessel wall imaging. Disagreement will be solved by consensus with involvement of a third expert.

SECONDARY OUTCOMES:
Quality of life related to the growth of UIA. | 5 years
  Evaluation of the quality of life (QOL) of untreated patients with UIA during the follow-up.
AWE variation patterns related to the growth of UIA. | 5 years
  Detection of other AWE variation patterns related to growth during the follow-up in order to improve the follow-up of UIA patients
Clinical, genetics or biological factors related to the growth of UIA. | 5 years
  Clinical, genetic (blood serum level of circulating ANGPTL6) and biological (plasma factors as circulating ANGPTL6 levels, metalloproteinase…) features recorded.
Incidence of growth of UIA. | 5 years
  Incidence of growth, stratified by clinical, genetics or biological features.
Incidence of IA rupture | 5 years
  Incidence of IA rupture, stratified by clinical, genetics or biological features.
quality of life patients related to the growth of UIA. | 5 years
  Completion of standardized EQ5D questionnaire to measure quality of life patients
Construction of an automatized tool of AWE pattern | 5 years
  Construction and evaluation of an automatized tool of AWE patterns, as compared to the visual analysis of experts, in the form of a decision-making tool.

CONTACTS AND LOCATIONS:
Overall Officials: Romain BOURCIER, MD, Principal Investigator — Nantes University Hospital
Locations (20):
- France (18):
  - Clairval's Hospital, Marseille, Bouches-du-Rhône
  - Brest University Hospital, Brest, Finistère
  - Bordeaux University Hospital, Bordeaux, Gironde
  - Toulouse University Hospital, Toulouse, Haute-Garonne
  - Limoges University Hospital, Limoges, Haute-Vienne
  - Rennes University Hospital, Rennes, Ille-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Angers University Hospital, Angers, Maine Et Loire
  - Reims University Hospital, Reims, Marne
  - Nancy University Hospital, Nancy, Meurthe-et-Moselle
  - Rouen University Hospital, Rouen, Seine-Maritime
  - Amiens University Hospital, Amiens, Somme
  - Creteil University Hospital, Créteil, Val-de-Marne
  - AP-HP La Pitié-Salpêtrière Hospital, Paris
  - AP-HP Le Kremlin Bicêtre Hospital, Paris
  - Rostchild Foundation Hospital, Paris
  - Ste Anne's Hospital, Paris, Île-de-France Region
- UMC Utrecht, Utrecht, Netherlands
- InselHospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided